CLINICAL TRIAL: NCT03440853
Title: Technology Assisted Stepped Collaborative Care Intervention (TASCCI) to Improve Patient-centered Outcomes in Hemodialysis Patients
Brief Title: Technology Assisted Stepped Collaborative Care Intervention
Acronym: TASCCI
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: University of Pittsburgh (Other)
Collaborators: National Institute of Diabetes and Digestive and Kidney Diseases (NIDDK) (NIH); University of New Mexico (Other)
Responsible Party: Principal Investigator, Manisha Jhamb, Associate Professor of Medicine, University of Pittsburgh
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: PRO17070630; 1R01DK114085-01 (NIH)
Record Dates: First submitted 2018-01-31; First posted 2018-02-22 (Actual); Last update posted 2022-07-11 (Actual); Status verified 2022-07

CONDITIONS: End-Stage Renal Disease; Hemodialysis
MeSH Terms: conditions — Kidney Failure, Chronic

STUDY DESIGN:
Intervention Model Description: Patients will be randomized 1:1 to TASCCI or technology-delivered health education and undergo a 12-week intervention. Psychological and clinical outcomes will be collected at baseline, post intervention, 6 and 12 months.
Who Masked: Outcomes Assessor
Masking Description: Patient reported outcomes will be administered centrally by blinded interviewers using computer-assisted telephone interviewing (CATI).
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- TASCCI (Experimental): Patients randomized to TASCCI will receive a stepped-care approach of pharmaco and/or behavioral therapy for 12 weeks. The intervention will target 1 or more symptoms based on patients' report of clinical levels of each symptom and patient preference.
  Interventions: Behavioral: TASCCI
- Technology Delivered Health Education (Other): Patients randomized to the Technology Delivered Health Education Intervention health education group will receive technology delivered health education material on topics relevant to dialysis.
  Interventions: Other: Technology Delivered Health Education Intervention

INTERVENTIONS:
Behavioral: TASCCI — TASCCI is a stepped-care collaborative care approach of pharmaco- and/or behavioral-therapy for a 12 week period. The intervention will target 1 or more symptoms based on patients' report of clinical levels of each symptom and patient preference. A trained behavioral therapist will deliver weekly video conferencing sessions during dialysis treatment.
  Arms: TASCCI
Other: Technology Delivered Health Education Intervention — The Technology Delivered Health Education Intervention will deliver weekly video conferencing sessions to deliver online educational material from the National Kidney Foundation. These sessions will be delivered by a care coordinator.
  Arms: Technology Delivered Health Education

SUMMARY:
This study evaluates a collaborative care intervention in reducing depression, fatigue and pain symptoms and improving health related quality of life in hemodialysis patients. Half of participants will receive the collaborative care intervention, while the other half will receive technology delivered health education information.

DETAILED DESCRIPTION:
End-stage renal disease patients on hemodialysis experience substantial symptom burden with fatigue, pain and depression among the most debilitating and existing as symptom clusters. These symptom clusters can exacerbate one another, and are independent and strong predictors of poor health-related quality of life in hemodialysis patients. This study will look at the effect of a 12 week stepped care intervention on changes in depression, pain or fatigue and health related quality of life.

ELIGIBILITY:
Inclusion Criteria:

1. 18 years or older
2. undergoing thrice-weekly maintenance hemodialysis for > 3 months
3. English speaking
4. able to provide informed consent
5. no evidence of thought disorder, delusions or active suicidal ideation

Exclusion Criteria:

1. thought disorder, delusions or active suicidal ideation
2. active substance abuse
3. too ill or cognitively impaired to participate based on clinicians' judgment
4. anticipated life expectancy of less than 1 year
5. unable or unwilling to adhere to study protocol
6. participating in another clinical trial or taking an investigational drug
7. scheduled for living donor kidney transplant within next 6 months
8. relocating to another dialysis unit within 6 months

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 160 (Actual)
Dates: Start 2018-03-28 (Actual); Primary Completion 2022-04-29 (Actual); Study Completion 2022-06-30 (Actual)

PRIMARY OUTCOMES:
Change in depression from baseline to 12 weeks | Baseline and Post 12 week intervention
  Depressive symptoms will be measured using the Beck Depression Inventory-II
Change in pain from baseline to 12 weeks | Baseline and Post 12 week intervention
  Pain symptoms will be measured using the Brief Pain Inventory
Change in fatigue from baseline to 12 weeks | Baseline and Post 12 week intervention
  Fatigue symptoms will be measured using the FACIT-F

SECONDARY OUTCOMES:
Change in adherence to medications | Baseline, 3 month, 6 month, 12 month
  Adherence will be measured using the Medication Adherence Questionnaire (MAQ) Morisky Green Levine
Change in adherence to fluid restriction | Baseline, 3 month, 6 month, 12 month
  Fluid restriction adherence will be determined by inter-dialytic weight gain percentage (of post dialysis weight over preceding 1 month) obtained by reviewing dialysis records. Those with IDWG% >3.5% will be classified as non-adherent
Change in adherence to hemodialysis treatments | Baseline and Post 12 week intervention
  Non-adherence with dialysis will be defined by the percentage of all dialysis sessions skipped and/or requested by the patient to be shortened by ≥ 10 minutes over the 12 week intervention period.

OTHER OUTCOMES:
To explore effect of TASCCI (hs-CRP, IL-6, IL-10 and TNF-α) on biomarkers of inflammation | Baseline and Post 12 week intervention, 6 month
  Effect of intervention on biomarkers of inflammation be measured by improvements in inflammatory cytokines.

CONTACTS AND LOCATIONS:
Overall Officials: Manisha Jhamb, MD, Principal Investigator — University of Pittsburgh
Locations (1):
- University of Pittsburgh, Pittsburgh, Pennsylvania, United States

REFERENCES:
- [Derived] Jhamb M, Steel JL, Yabes JG, Roumelioti ME, Erickson S, Devaraj SM, Vowles KE, Vodovotz Y, Beach S, Weisbord SD, Rollman BL, Unruh M. Effects of Technology Assisted Stepped Collaborative Care Intervention to Improve Symptoms in Patients Undergoing Hemodialysis: The TACcare Randomized Clinical Trial. JAMA Intern Med. 2023 Aug 1;183(8):795-805. doi: 10.1001/jamainternmed.2023.2215. PMID 37338898